CLINICAL TRIAL: NCT04307823
Title: Effects of Respiratory Muscles Training on Cardiopulmonary Parameters and Quality of Life in Patients With Dilated Cardiomyopathy
Brief Title: Respiratory Muscles Training in Patients With Dilated Cardiomyopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00596 Hanifa Suleman
Record Dates: First submitted 2020-03-02; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Dilated Cardiomyopathy
Keywords: Bruce protocol; Congestive heart failure; Dilated cardiomyopathy; Incentive spirometry; Slow breathing training
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill training group (Active Comparator): Treadmill training according to American College of Sports Medicine's guidelines
  Interventions: Other: Treadmill training
- Treadmill protocol and respiratory training group (Experimental): Treadmill training, slow breathing training and incentive spirometry
  Interventions: Other: Treadmill protocol and Respiratory training

INTERVENTIONS:
Other: Treadmill training — 3 days per week, starting at shorter duration 5-20min and progressed to 30- 40mins.
  Training% or Intensity was kept 40-70%,
  Training Heart Rate (HR) was calculated through formula:
  HR max HR rest*Ex intensity + HR rest Rate of Perceived Exertion (RPE) 9-14 ON 6 -20 RPE scale The session was terminated if sustained ventricular arrhythmia, symptomatic drop in blood pressure, ST elevation, or development of severe symptoms
  Arms: Treadmill training group
Other: Treadmill protocol and Respiratory training — Treadmill protocol
  Spirometry:
  Volumetric exercises, using incentive Spirometer 10-15 repetitions
  Slow breathing training:
  5 minutes: spontaneous breathing, 4 minutes: controlled breathing (15 breaths/min) 4 minutes of controlled breathing (6 breaths/min) Treatment provided for 3 days in a week for a period of 4 weeks
  Arms: Treadmill protocol and respiratory training group

SUMMARY:
The aim of this study was to determine the effects of respiratory muscles training on cardiopulmonary parameters and quality of life in patients with dilated cardiomyopathy (DCM). It was a randomized control trial conducted on the calculated sample size of 22 patients divided into 2 groups. Study was conducted at Shifa International Hospital Islamabad. Clinically stable, diagnosed cases of DCM aged 30 to 60 years were included in the study. Outcomes of study were ejection fraction, Left ventricular (LV) End systolic dimensions, LV End diastolic dimension, lung volumes and capacities and quality of life. Data was analyzed on Statistical Package for the Social Sciences (SPSS) version 21.

.

DETAILED DESCRIPTION:
Dilated cardiomyopathy is the most common type of heart failure and primary source of heart replacement globally. It is characterized by poor left ventricular function,enlargement of left ventricle and systolic dysfunction. The underlying cause of DCM in adults is usually coronary artery disease, but other causes include inflammatory heart disease, myocardial toxins, and genetic defects; approximately 30% to 35% of patients are reported to have a genetic form of dilated cardiomyopathy. Most common sign and symptoms of dilated cardiomyopathy are ankle swelling, dyspnea, fatigue, elevated jugular venous pressure elevated, pulmonary rales due to reduced cardiac function with low output and elevated intra cardiac pressures. Other sign and symptoms chest pain due to reduced coronary blood flow, palpitation, syncope and sudden cardiac death. There is reduced exercise tolerance with fatigue and dyspnea, contributing to poor prognosis and quality of life.

Chronic heart failure (CHF) patients have limited capacity to exercise and have impairments in breathing function.Respiratory muscle weakness is a part of the underlying cause for exercise intolerance in patients with heart failure with reduced ejection fraction.

Pharmacological and non pharmacological management is directed to reduce clinical sign and symptoms and control of disease progression and complications like sudden cardiac arrest. Physical rehabilitation is beneficial, effective and safe for functional limitation of DCM patients. A modified Bruce protocol is usually used to gradually increase exercise intensity in cardiac rehabilitation programs for patients with cardiomyopathy. Bruce protocol was used to observe fluctuations in heart rate through a quick increase of exercise intensity for a short period of time. Some patients are able to exercise with higher intensity safely, but many patients reported difficulties on treadmill exercise. This becomes even more difficult when the intensity of the treadmill exercise is increased.

Various studies have demonstrated the effects of exercise as well as inspiratory muscle training for improvement in patients with CHF and have considered it an important component of cardiac rehabilitation. Respiratory muscles training is commonly performed using inspiratory resistance devices but studies have proven that incentive spirometry could be an interesting alternative for clinical use for the cases where there is difficult to acquire the devices. Slow breathing treatment is safe and induces favourable effects in cardiopulmonary parameters, decreases rate of dyspnea, improves exercise performance and increases respiratory muscles and function. Deeper and slow breathing involves the use of diaphragm that is activated during slow breathing and does not increase respiratory workload.Respiratory muscles training is safe and improves physiologic parameters including an increase in oxygen saturation and improved exercise capacity, leading to an improvement in health status.

This study is intended to observed the overall effect of respiratory muscles training including slow breathing and incentive spirometry along with treadmill training according to bruce protocol for improvement in their ejection fraction, left ventricular dimensions , pulmonary function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of DCM
* New York Heart Association class (II)
* Clinically stable patients for at least (3) months
* Ejection Fraction (25 - 40%)

Exclusion Criteria:

* Recent myocardial infarction, exercise induced angina and Syncope,
* Atrioventricular valve disease, selected for heart transplant
* Uncontrolled hypertension.
* Uncontrolled diabetes.
* Significant pulmonary disease. Intellectual, neurological or musculoskeletal abnormalities.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Ejection fraction | After 4 weeks of intervention
  Ejection fraction calculated through echocardiography
LV End systolic dimension | After 4 weeks of intervention
  LV End systolic dimension calculated through echocardiography
LV End diastolic dimension | After 4 weeks of intervention
  LV End diastolic dimension calculated through echocardiography

SECONDARY OUTCOMES:
Memorial symptom assessment scale - Heart failure | After 4 weeks of intervention
  Memorial symptom assessment scale for heart failure patients (MSAS-HF) is a patient-rated instrument to assess the quality of life of heart failure patients. It scores 32 symptoms including 26 physical symptoms of distress and 6 psychological symptoms are recorded.
  Distress is rated on a 5 point scale each symptom is scored from 0 to 4 ranging from "no symptom" to "very much." If the symptom is not present, a value of zero is assigned.
  Frequency of psychological symptoms is scored as 1-rarely, 2- occasionally, 3-frequently, and 4- almost constantly.
  The symptom scores are combined into various sub-scales scores including the psychological sub-scale score, physical sub-scale, global distress index and total MSAS score. The mean score in each category is calculated with higher scores indicating poor quality of life.
Forced Expiratory volume 1(FEV1) | After 4 weeks of intervention
  Forced Expiratory volume 1(FEV1) measured through digital spirometer. If the value of FEV1 is within 80% of the reference value, the results are considered normal.
Forced Vital capacity(FVC) | After 4 weeks of intervention
  Forced Vital capacity(FVC) measured through digital spirometer. If the value of FVC is within 80% of the reference value, the results are considered normal.
FEV1/FVC | After 4 weeks of intervention
  FEV1/FVC measured through digital spirometer. The normal value for the FEV1/FVC ratio is 70% (and 65% in persons older than age 65).
Peak Expiratory Flow Rate (PEFR) | After 4 weeks of intervention
  Peak Expiratory Flow Rate (PEFR) measured through digital spirometer. Three zones of measurement are commonly used to interpret peak flow rates. Normal value of PEFR is (80-100%). Green zone indicates 80 to 100 percent of the usual or normal peak flow reading, yellow zone indicates 50 to 79 percent of the usual or normal peak flow readings, and red zone indicates less than 50 percent of the usual or normal peak flow readings.

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ziaeian B, Fonarow GC. Epidemiology and aetiology of heart failure. Nat Rev Cardiol. 2016 Jun;13(6):368-78. doi: 10.1038/nrcardio.2016.25. Epub 2016 Mar 3. PMID 26935038
- [Background] Russo MA, Santarelli DM, O'Rourke D. The physiological effects of slow breathing in the healthy human. Breathe (Sheff). 2017 Dec;13(4):298-309. doi: 10.1183/20734735.009817. PMID 29209423
- [Background] Drozdz T, Bilo G, Debicka-Dabrowska D, Klocek M, Malfatto G, Kielbasa G, Styczkiewicz K, Bednarek A, Czarnecka D, Parati G, Kawecka-Jaszcz K. Blood pressure changes in patients with chronic heart failure undergoing slow breathing training. Blood Press. 2016;25(1):4-10. doi: 10.3109/08037051.2016.1099800. Epub 2015 Oct 29. PMID 26513698
- [Background] Wasserstrum Y, Barbarova I, Lotan D, Kuperstein R, Shechter M, Freimark D, Segal G, Klempfner R, Arad M. Efficacy and safety of exercise rehabilitation in patients with hypertrophic cardiomyopathy. J Cardiol. 2019 Nov;74(5):466-472. doi: 10.1016/j.jjcc.2019.04.013. Epub 2019 Jun 22. PMID 31235420
- [Background] Gomes-Neto M, Duraes AR, Conceicao LSR, Roever L, Silva CM, Alves IGN, Ellingsen O, Carvalho VO. Effect of combined aerobic and resistance training on peak oxygen consumption, muscle strength and health-related quality of life in patients with heart failure with reduced left ventricular ejection fraction: a systematic review and meta-analysis. Int J Cardiol. 2019 Oct 15;293:165-175. doi: 10.1016/j.ijcard.2019.02.050. Epub 2019 Jun 24. PMID 31345646
- [Background] Lachowska K, Bellwon J, Morys J, Gruchala M, Hering D. Slow breathing improves cardiovascular reactivity to mental stress and health-related quality of life in heart failure patients with reduced ejection fraction. Cardiol J. 2020;27(6):772-779. doi: 10.5603/CJ.a2019.0002. Epub 2019 Jan 30. PMID 30697682
- [Background] Neto MG, Martinez BP, Conceicao CS, Silva PE, Carvalho VO. Combined Exercise and Inspiratory Muscle Training in Patients With Heart Failure: A SYSTEMATIC REVIEW AND META-ANALYSIS. J Cardiopulm Rehabil Prev. 2016 Nov/Dec;36(6):395-401. doi: 10.1097/HCR.0000000000000184. PMID 27182763
- [Background] Leggio M, Fusco A, Loreti C, Limongelli G, Bendini MG, Mazza A, Coraci D, Padua L. Effects of exercise training in heart failure with preserved ejection fraction: an updated systematic literature review. Heart Fail Rev. 2020 Sep;25(5):703-711. doi: 10.1007/s10741-019-09841-x. PMID 31399956